CLINICAL TRIAL: NCT01722643
Title: Incentives, Cognitive Training and Internet Therapy for Teens With Poorly Controlled Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Catherine Stanger, Associate Professor, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23559; 1DP3HD076602-01 (NIH)
Record Dates: First submitted 2012-10-19; First posted 2012-11-07 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MAxIM (Experimental): This new intervention, called MAxIM (MotivAtion, Incentives, Memory) uses: 1) motivation enhancement therapy (MET) (an existing evidence-based treatment for adolescent with diabetes) supplemented with cognitive behavior therapy (CBT) to enhance behavior change; 2) financial incentives for daily blood glucose testing and parental monitoring to provide frequent positive feedback; and 3) working memory training (WMT), a method for strengthening specific cognitive processes that support decision-making and future orientation. The interventions will be delivered to families at home via the internet.
  Interventions: Behavioral: MAxIM
- Usual Care (Active Comparator): Usual Care reflects the standard treatment currently provided at the Children's Hospital at Dartmouth. Teens will be followed by their treating endocrinologist and receive the following standard services as part of that treatment-quarterly outpatient clinic visits, including an interval medical history and physical examination; routine laboratory assessment; review of glycemic control, medication adjustment, medical nutrition therapy, and diabetes self-management education; telephone consultations with a nurse/certified diabetes educator in their treating clinic are available as often as necessary between clinic visits.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: MAxIM — This new intervention, called MAxIM (MotivAtion, Incentives, Memory) uses: 1) motivation enhancement therapy (MET) (an existing evidence-based treatment for adolescent with diabetes) supplemented with cognitive behavior therapy (CBT) to enhance behavior change; 2) financial incentives for daily blood glucose testing and parental monitoring to provide frequent positive feedback; and 3) working memory training (WMT), a method for strengthening specific cognitive processes that support decision-making and future orientation. The interventions will be delivered to families at home via the internet.
  Arms: MAxIM
Behavioral: Usual Care — Usual Care reflects the standard treatment currently provided at the Children's Hospital at Dartmouth. Teens will be followed by their treating endocrinologist and receive the following standard services as part of that treatment-quarterly outpatient clinic visits, including an interval medical history and physical examination; routine laboratory assessment; review of glycemic control, medication adjustment, medical nutrition therapy, and diabetes self-management education; telephone consultations with a nurse/certified diabetes educator in their treating clinic are available as often as necessary between clinic visits.
  Arms: Usual Care

SUMMARY:
The overall goal of this project is to develop a novel family friendly intervention that will help teens with poor metabolic control of their type 1 diabetes increase and sustain daily self monitoring of blood glucose and lower HbA1c. This is important because poor metabolic control has long-term health implications. This project will provide important information regarding new effective ways to improve outcomes among teens with poorly controlled type 1 diabetes.

Primary hypotheses are that the intervention, MAxIM, will: (1) help teens improve and maintain glucose control, and (2) improve decision making (improve executive function and reduce delay discounting), which will predict treatment outcome.

DETAILED DESCRIPTION:
Type 1 diabetes in adolescents is a significant medical condition associated with high economic costs and increased mortality, and its incidence is increasing. Unfortunately, adolescents show poorer adherence to self monitoring of blood glucose (SMBG) recommendations and poorer metabolic control than adults. Although some individual and family-based interventions have shown promise in improving metabolic control, there is a critical need to develop more effective interventions. The overall goal of this DP3 project is to develop a new innovative intervention that targets decision making to help teens with poor diabetic metabolic control increase the frequency of SMBG and improve HbA1c. The target population will be teens aged 13-17 with type 1 diabetes and HbA1c >8%. Based on our prior work and a conceptual model, the proposed study will develop and pilot test a novel, multifaceted, developmentally appropriate intervention aimed at improving adolescent decision making. An integrated set of components target adolescents' need for frequent positive feedback, improved future orientation, and motivational support. While past research indicates that behavioral interventions are frequently more successful when they include multiple elements, no previous intervention has combined multiple empirically-based components that target key decision making levers in one intervention. This new intervention, called MAxIM (MotivAtion, Incentives, Memory) uses: 1) motivation enhancement therapy (MET) (an existing evidence-based treatment for adolescent with diabetes) supplemented with cognitive behavior therapy (CBT) to enhance behavior change; 2) financial incentives for daily blood glucose testing and parental monitoring to provide frequent positive feedback; and 3) working memory training (WMT), an efficacious method for strengthening specific cognitive processes that support decision-making and future orientation. The interventions will be delivered to families at home via the internet to increase the reach of the intervention to families living distant from their treating endocrinologist. MAxIM will be teen and parent friendly and designed to increase engagement and compliance with the intervention. Primary hypotheses are that MAxIM will: (1) help teens improve and maintain glucose control, and (2) improve decision making (improve executive function and reduce delay discounting), which will predict treatment outcome. The unique set of interventions holds promise for improving adherence by affecting multiple basic mechanisms that determine poor decision making. The project will develop a novel, highly transportable, home based intervention designed to maximize and sustain HbA1c reductions and SMBG frequency over time in adolescents. Innovations include the targeting of multiple levers specific to adolescent decision making, use of technology to deliver the intervention to families at home, and testing cognitive predictors of treatment outcome for teens with diabetes. Successful achievement of this study's aims will bring the field closer to a cost effective, long-lasting intervention to improve outcomes among these high-risk youth.

ELIGIBILITY:
Inclusion Criteria:

* 13-17 years old
* Diagnosis of type 1 diabetes
* Average HbA1c > or = to 8% for the past 6 months (mean of two values)
* Most recent HbA1c is > or = to 8%
* Duration of disease is > 18 months
* Teen must live at home
* Family must have broadband internet in the home

Exclusion Criteria:

* Pregnancy/breast feeding
* Active psychosis
* Severe medical or psychiatric illness that will limit participation

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2014-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Stanger, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth College, Hanover, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crochiere RJ, Hughes Lansing A, Carracher A, Vaid E, Stanger C. Attentional bias to diabetes cues mediates disease management improvements in a pilot randomized controlled trial for adolescents with type 1 diabetes. J Health Psychol. 2021 Dec;26(14):2699-2710. doi: 10.1177/1359105320926535. Epub 2020 Jun 7. PMID 32508201
- [Derived] Stanger C, Lansing AH, Scherer E, Budney A, Christiano AS, Casella SJ. A Web-Delivered Multicomponent Intervention for Adolescents with Poorly Controlled Type 1 Diabetes: A Pilot Randomized Controlled Trial. Ann Behav Med. 2018 Nov 12;52(12):1010-1022. doi: 10.1093/abm/kay005. PMID 30418521

RESULTS

PARTICIPANT FLOW:
Groups:
- MAxIM: This intervention, called MAxIM (MotivAtion, Incentives, Memory) uses: 1) motivation enhancement therapy (MET) (an existing evidence-based treatment for adolescent with diabetes) supplemented with cognitive behavior therapy (CBT) to enhance behavior change; 2) financial incentives for daily blood glucose testing and parental monitoring to provide frequent positive feedback; and 3) working memory training (WMT), a method for strengthening specific cognitive processes that support decision-making and future orientation. The interventions will be delivered to families at home via the internet.
- Usual Care: Usual Care reflects the standard treatment currently provided for type 1 diabetes. Teens will be followed by their treating endocrinologist and receive standard services as part of that treatment-quarterly outpatient clinic visits, including an interval medical history and physical examination; routine laboratory assessment; review of glycemic control, medication adjustment, medical nutrition therapy, and diabetes self-management education; telephone consultations with a nurse/certified diabetes educator in their treating clinic are available as often as necessary between clinic visits.
Period: Overall Study
Arm/Group | MAxIM | Usual Care
Started | 30 | 31
Completed | 30 | 30
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MAxIM | Usual Care | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.2 (1.4) | 14.9 (1.5) | 15.1 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 19 | 16 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 29 | 31 | 60
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 30 | 30 | 60
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 31 | 61
HbA1c [Mean (Standard Deviation); unit: percentage glycated hemoglobin] | 9.1 (1.0) | 9.2 (0.9) | 9.1 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c at 12 Months
Description: Glycated hemoglobin test (HbA1c) measures the non-enzymatic glycation status of hemoglobin expressed in percentage points. Analyses control for pump status, diabetes duration and baseline HbA1c
Time Frame: 12 months following enrollment
Measure: Least Squares Mean (Standard Error); unit: percentage glycated hemoglobin
Arm/Group | MAxIM | Usual Care
Number analyzed (Participants) | 30 | 30
percentage glycated hemoglobin | 8.73 (0.18) | 9.29 (0.18)

2. Secondary Outcome: Daily Frequency of Self Monitoring of Blood Glucose Checks 12 Months Following Enrollment
Description: Participants will use a glucometer to self-monitor blood glucose daily. Readings from the glucometer will be uploaded at each session and at the follow up visits. The glucometer records the blood glucose level as well as a date/time stamp over a 90 day period. To assess the daily testing frequency, the total number of blood glucose tests a day during the 14 days prior to each assessment will be recorded from the study provided glucometer.
Time Frame: 12 months following enrollment
Population: 1 participant in the MaxIM arm and 1 participant in the Usual Care arm did not provide meter data at 12 months so do not have data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: readings per day
Arm/Group | MAxIM | Usual Care
Number analyzed (Participants) | 29 | 29
readings per day | 4.75 (.33) | 3.56 (.33)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events were collected at each assessment through 12 months via the Health Services Utilization form (Huang, E. S., O'Grady, M., Basu, A., Winn, A., John, P., Lee, J., ... & Wysocki, T. (2010). The cost-effectiveness of continuous glucose monitoring in type 1 diabetes. Diabetes care, 33(6), 1269-1274.)
Arm/Group | MAxIM | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/30 | 3/31
Other Adverse Events (participants affected / at risk) | 1/30 | 1/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAxIM (N=30) | Usual Care (N=31)
ER visit with or without hospitalization for low blood sugar (Endocrine disorders) | 0 (0) | 2 (3)
ER visit with or without hospitalization for high blood sugar (Endocrine disorders) | 1 (1) | 2 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MAxIM (N=30) | Usual Care (N=31)
Severe low blood sugar event requiring assistance to treat (Endocrine disorders) | 1 (28) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No